CLINICAL TRIAL: NCT06651099
Title: A Multicenter Trial-based Economic Evaluation of a Mobile Health Intervention for Individuals With Chronic Non-specific Low Back Pain: Randomized Controlled Trial (eBack Trial)
Brief Title: Trial-based Economic Evaluation of a Mobile Health Intervention for Individuals With Chronic Non-specific Low Back Pain
Acronym: eBack
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: VU University of Amsterdam (Other); Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Prof. Rodrigo Luiz Carregaro, Prof. Dr., University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6.674.643
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: Back pain; Mobile health; Economic evaluation; Exercise therapy; Self-management
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: Multicenter trial-based economic evaluation comparing mhealth intervention versus a conventional exercise therapy intervention alone. All participants will be randomly assigned to one of two groups: 1) blended mhealth intervention (mhG) or 2) conventional exercise therapy delivered by a booklet (beG).
Who Masked: Outcomes Assessor
Masking Description: Blinding the therapists will not be possible due to the nature of the interventions. Because outcomes are self-reported, blinding participants to the intervention will also not be possible. However, an assessor who will be unaware of the group allocation will perform the data collection. The researcher responsible for the statistical analysis will also be blinded to the group allocation (i.e. they will receive the data sheet with the groups/individuals coded numerically).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mhealth application (experimental group) (Experimental): The mhealth intervention group will be instructed to perform the exercises twice a week for 8 weeks, lasting approximately 30 minutes per session. Participants will be instructed to watch the health education content (e.g., short videos, infographics) and exercise videos provided by the app, and to take breaks during each session. Guidance will be provided during the intervention and weekly monitoring by a physiotherapist by messaging or telephone calls. In the first week of the intervention there will be two face-to-face sessions supervised by the physiotherapist to familiarize the participants with the mobile application and provide instructions on the intervention. A further face-to-face session will take place half-way the intervention, to monitor the participants.
  Interventions: Other: mhealth application
- Conventional booklet exercise (comparator group) (Active Comparator): After the assessment, all participants will receive a printed booklet containing a description and recommendations for carrying out the exercise program at home, which will be characterized by general exercises (i.e., strengthening, mobilization). The individuals will be instructed to perform the exercises twice a week for 8 weeks, following the same duration on the experimental group. Participants will be monitored and supervised by another physiotherapist via messaging app or telephone calls, following the same procedures reported in the experimental group. In the first week of the intervention there will be two face-to-face sessions supervised by a physiotherapist to familiarize the participants with the exercises and explain the booklet, and provide instructions on the intervention. A further face-to-face session will take place half-way the intervention, to monitor the participants.
  Interventions: Other: Conventional exercise therapy

INTERVENTIONS:
Other: mhealth application — Individuals enrolled in the mhealth intervention will receive tailored content will include exercises focused on mobility, flexibility, core stabilization, and strengthening. Additionally, the mobile application will provide educational material on pain and health, covering topics such as the neurophysiology of pain, the multidimensional nature of low back pain, myths and facts about the condition, the importance of sleep, and stress management, which will include relaxation techniques and mindfulness. All content will be evidence-based, using clinical guidelines, systematic reviews and other high-quality studies to support inclusion in the mobile application. The intervention will be supervised by a physiotherapist, remotely via messaging or telephone calls.
  Arms: mhealth application (experimental group)
Other: Conventional exercise therapy — Participants in this intervention will receive a printed booklet containing a description and recommendations for carrying out an exercise program at home, which will be characterized by general exercises (such as strengthening, mobilization). The intervention will be supervised by a physiotherapist, remotely via messaging or telephone calls.
  Arms: Conventional booklet exercise (comparator group)

SUMMARY:
The aim of this trial is to assess the effectiveness and cost-effectiveness of a supervised and more personalised mhealth intervention compared with conventional exercise therapy in people with chronic non-specific low back pain.

DETAILED DESCRIPTION:
Background: Chronic non-specific low back pain (CNLBP) is a prevalent and costly condition that encourages research into self-management strategies. Mobile health (mhealth) applications are promising interventions, but current evidence on their effectiveness is still conflicting. The aim is to investigate the (cost-)effectiveness of a supervised and personalized mhealth intervention, compared with conventional exercise therapy in individuals with CNLBP. Methods: A multicentre trial-based economic evaluation was designed to compare a mhealth intervention with conventional exercise. Participants will be recruited from two physical therapy rehabilitation clinics located within the participating centres. Adults aged between 18 and 59 years and with self-reported LBP >12 weeks will be included. Following the collection of baseline data, participants will be randomly assigned to one of two groups using a permuted block randomization: 1) mhealth; 2) Conventional exercise delivered through a booklet. Outcome assessments will be conducted following randomisation at five distinct time points, resulting in a total follow-up period of 12 months. The primary clinical outcome is disability (Roland-Morris Disability Questionnaire), while secondary outcomes include pain (NRS), utility (EQ5D5L), fears and beliefs (FABQ), self-efficacy (PSEQ), and global perceived effect. A sample size of 146 participants was estimated (73 allocated to each group) in order to detect a 2-point between-groups difference on disability. A cost-effectiveness study will be conducted alongside the trial, comparing the two interventions in terms of costs and clinical outcomes. Discussion: While mhealth applications show promise as interventions for people with LBP, there is still a gap regarding the type of delivery and personalisation strategies. This study investigates whether the implementation of stratified and tailored care within a mobile application, based on patient-reported outcome measures and supervised by a physiotherapist, is (cost)effective.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 59 years;
* Self-reported low back pain for more than 12 consecutive weeks prior to the study, with pain intensity ≥4 in the numerical rating scale (NRS);
* Not having participated in physiotherapy sessions for treatment of low back pain for at least 6 months prior to the start of the study;
* Having a smartphone with internet access;
* Self-management activation classified as Level 2 or higher (i.e., classifications of low, medium and high knowledge about self-management), according to the Patient Activation Measure (PAM) questionnaire.

Exclusion Criteria:

* History of spinal trauma or fracture;
* Diagnosis of spinal osteoarthritis, fibromyalgia, or rheumatic diseases; 3) Referred pain (from viscera, appendicitis, abdominal and pelvic pain);
* Previous spinal surgery;
* Presence of red flags, signs and/or symptoms of neurological impairment and/or pain radiating below the knee;
* Pregnancy.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Disability score as assessed by the Roland-Morris Disability Questionnaire | From enrollment to the end of treatment (around eight to ten weeks from baseline), and follow-up moments: follow-up 1 (26 weeks after baseline); follow-up 2 (39 weeks after baseline), and follow-up 3 (52 weeks after baseline)
  Disability will be the primary clinical outcome and will be measured using the Brazilian-portuguese validated version of the Roland-Morris Disability Questionnaire (RMDQ). The questionnaire consists of 24 items with 0=no and 1=yes, and the total score ranges from zero (no disability) to 24 (severe disability).

SECONDARY OUTCOMES:
Pain intensity as measured using the Numerical Rating Scale (NRS) | From enrollment to the end of treatment (around eight to ten weeks from baseline), and follow-up moments: follow-up 1 (26 weeks after baseline); follow-up 2 (39 weeks after baseline), and follow-up 3 (52 weeks after baseline)
  Pain intensity will be measured using the Numerical Rating Scale (NRS). This scale is characterized by a line with unit scores ranging from 0 to 10, where zero corresponds to no pain and ten corresponds to the worst pain ever experienced. Participants will be instructed to mark a number on the line, representing the pain intensity in the last week
Health-related quality of life (Utility) as measured by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire | From enrollment to the end of treatment (around eight to ten weeks from baseline), and follow-up moments: follow-up 1 (26 weeks after baseline); follow-up 2 (39 weeks after baseline), and follow-up 3 (52 weeks after baseline)
  The Brazilian-portuguese version of the EQ-5D-5L questionnaire available at Euroqol will be used to assess participants' utility based on five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels (i.e., no problems, slight problems, moderate problems, severe problems, and extreme problems). The scores range from 0 (the value of a health status equivalent to death) to 1 (the value of full health), with higher scores indicating greater health utility.
Fear and beliefs as measured by the Fear Avoidance Beliefs Questionnaire | From enrollment to the end of treatment (around eight to ten weeks from baseline), and follow-up moments: follow-up 1 (26 weeks after baseline); follow-up 2 (39 weeks after baseline), and follow-up 3 (52 weeks after baseline)
  Fear and beliefs will be assessed using the validated Brazilian version of the FAB-Q (Fear Avoidance Beliefs Questionnaire). The FABQ consists of 16 self-report items, divided into two subscales: FABQ-Work, which addresses individuals' fears and beliefs in relation to work, and FABQ-Phys, which addresses their fears and beliefs in relation to physical activities. Each item is assessed on a seven-point Likert scale, ranging from 0 (completely disagree) to 6 (completely agree).
Self-efficacy as measured by the Self-Efficacy Questionnaire (PSEQ) | From enrollment to the end of treatment (around eight to ten weeks from baseline), and follow-up moments: follow-up 1 (26 weeks after baseline); follow-up 2 (39 weeks after baseline), and follow-up 3 (52 weeks after baseline)
  Self-efficacy will be assessed using the the Pain Self-Efficacy Questionnaire (PSEQ), translated and validated for Brazilian Portuguese. The PSEQ is a 10-item questionnaire designed to assess the confidence of people with persistent pain in performing various activities, even in the presence of pain. Each item is scored on a 7-point numerical scale (scores from 0 to 6), where 0 means 'not at all confident' and 6 means 'completely confident'. The items assess self-efficacy for a range of functions, including housework, socialising, work, and pain management without medication and with medication. The total score is obtained by summing the scores of the 10 items, resulting in a value between 0 and 60. Higher scores indicate greater perceived self-efficacy.
Perceived recovery as measured by the Global Perceived Effect Scale | At the end of treatment (around eight to ten weeks from baseline), and follow-up moments: follow-up 1 (26 weeks after baseline); follow-up 2 (39 weeks after baseline), and follow-up 3 (52 weeks after baseline)
  Perceived recovery will be assessed at the end of the intervention period and follow-up moments using the Global Perceived Effect Scale (11-point scale), ranging from -5 ('much worse'), 0 ('no change') to 5 ('completely recovered')

OTHER OUTCOMES:
Quality-adjusted life years (QALY) | From enrollment to the end of treatment (around eight to ten weeks from baseline), and follow-up moments: follow-up 1 (26 weeks after baseline); follow-up 2 (39 weeks after baseline), and follow-up 3 (52 weeks after baseline)
  The QALY will be calculated from the utilities assessed at each of the 5 time points by the EQ-5D-5L questionnaire using the area under the curve method. In this approach, the average utility values between each two time points for each participant are multiplied by the corresponding time periods in weeks. The resulting values are then summed to obtain the total QALYs over the study period (12 months).
Cost-effectiveness | From enrollment to the end of treatment (around eight to ten weeks from baseline), and follow-up moments: follow-up 1 (26 weeks after baseline); follow-up 2 (39 weeks after baseline), and follow-up 3 (52 weeks after baseline)
  Cost outcomes will include healthcare costs (i.e., healthcare utilization costs and intervention costs) and total societal costs (i.e., healthcare utilization costs, intervention costs, informal care costs, and lost productivity costs). Incremental cost-effectiveness ratios (costs per clinical outcome) and cost-utility ratios (costs per QALY gained) will be calculated from the perspectives of the public health system and society.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo L Carregaro, PhD, Study Director — University of Brasilia; Fernanda Pasinato, PhD, Study Chair — University of Brasilia; Thomaz N Burke, PhD, Study Chair — Federal University of Mato Grosso
Locations (2):
- Brazil (2):
  - Universidade de Brasília, Ceilândia, Federal District
  - Federal University of Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Araujo Mota MA, Landolfi TB, de Melo Silva MC, de Melo Santana B, Ben AJ, van Dongen JM, Bosmans JE, Ostelo R, Burke TN, Pasinato F, Tottoli CR, Luiz Carregaro R. A multicenter trial-based economic evaluation of a mobile health intervention for individuals with chronic non-specific low back pain: randomized controlled trial protocol. BMC Musculoskelet Disord. 2025 Aug 23;26(1):814. doi: 10.1186/s12891-025-09118-5. PMID 40849470